CLINICAL TRIAL: NCT06038955
Title: Effect of Immersive Virtual Reality-based Cognitive Remediation in Patients With Mood Disorders or Psychosis Spectrum Disorders: a Randomized, Controlled, Double-blinded Trial
Brief Title: Effect of Immersive Virtual Reality-based Cognitive Remediation in Patients With Mood - or Psychosis Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry); University of Copenhagen (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kamilla Woznica Miskowiak, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-22004153; P-2022-411 (Other: Registry ID: Danish Data Protection Agency)
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-01

CONDITIONS: Bipolar Disorder; Depression; Psychotic Disorders; Cognitive Impairment; Schizophrenia; Schizotypal Disorder
Keywords: Cognition; Cognitive Impairment; Cognitive Remediation; Depression; Bipolar Disorder; Schizophrenia; Schizotypal Disorder; Psychotic Disorders; Virtual Reality
MeSH Terms: conditions — Bipolar Disorder; Depression; Psychotic Disorders; Cognitive Dysfunction; Schizophrenia; Schizotypal Personality Disorder

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blinded, parallel-group design
Who Masked: Participant, Outcomes Assessor
Masking Description: The study has a double-blinded design. Neither the participant nor the outcome-assessors will know whether the participant is receiving VR-based cognitive remediation or VR control treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality Based Cognitive Remediation (Experimental): The cognitive remediation program has a duration of four weeks and involves two weekly 1,5-hour virtual reality-based cognitive training sessions with a therapist accompanied by additional between-session virtual reality training at home and homework assignments consisting of cognitively challenging daily life tasks.
  Interventions: Behavioral: Virtual reality Based Cognitive Remediation
- Virtual reality control treatment (Sham Comparator): The control treatment program also has a duration of four weeks and involves one weekly 2-hour session with a therapist.
  Interventions: Behavioral: Virtual reality control training

INTERVENTIONS:
Behavioral: Virtual reality Based Cognitive Remediation — The main component of the intervention is a virtual reality training platform in 360° Oculus Quest 2-software in which participants train their cognitive abilities guided by the therapist. The platform includes four immersive daily-life scenarios in which patients have consistently reported that they often experience cognitive difficulties: (1) a kitchen scenario focusing on planning and cooking a meal, (2) a supermarket scenario focusing on grocery shopping, (3) a restaurant scenario focusing on remembering names and personal information and (4) an office scenario focusing on planning, initiating, and completing work assignments. The virtual reality training is supported by a psychoeducation program that focuses on application of learned cognitive strategies in daily life.
  Arms: Virtual reality Based Cognitive Remediation
Behavioral: Virtual reality control training — The virtual reality control training involves completing different virtual reality games that are available through the Oculus Quest games store.The chosen games involve no direct training of cognitive abilities such as planning skills og strategic learning, but merely involves simple reaction time and interaction with an entertaining environment that is meaningful to the participant and gives the impression of training cognitive skills.
  Arms: Virtual reality control treatment

SUMMARY:
The goal of this clinical trial is to investigate the effect of a four-weeks, intensive virtual reality (VR)-based cognitive remediation (training) programme involving simulated daily-life challenges on cognition and functional capacity in symptomatically stable patients with mood disorders (depression or bipolar disorder) or psychosis spectrum disorders (F20-F29; e.g. schizophrenia or schizotypal disorder).

The investigators hypothesize that VR-based cognitive remediation vs. a VR control treatment has a beneficial effect on cognition after four-weeks treatment completion (primary outcome assessement time) measured with a novel ecologically valid VR test of daily-life cognitive functions (The CAVIR test; primary outcome measure), a verbal learning and memory composite score based on a traditional neuropsychological test and a performance-based measure of daily functioning (secondary outcome measures). Finally, for exploratory purposes, the study will examine neuronal underpinnings of treatment effects, and effects on additional measures of cognition, functioning and self-ratings scales (tertiary outcomes).

DETAILED DESCRIPTION:
The current study will include outpatients with a mood disorders (unipolar - or bipolar disorder) in full or partial remission at the time of inclusion (score ≤ 14 on the Hamilton Depression or a psychosis spectrum disorders (F20-F29) that have been assessed to be relatively symptom stable by their treating clinician upon referral to the study. To accommodate for an approximately 20% drop-out rate from baseline to treatment completion (the primary outcome assessement time point), the investigators will recruit up to 66 participants (33 participants per intervention arm) to obtain complete data for minimum 54 participants (27 participants per arm).

Recruitment will be carried out through the outpatient Copenhagen Affective Disorder Clinic, the outpatient, early intervention clinics for psychotic disorders (OPUS), other mental health centres in the Capital Region of Denmark, and through advertisements on relevant websites.

After inclusion, the baseline assessements are scheduled and completed over two days, one to five days apart. On day 1, the participant is assessed with the virtual cognition test (the CAVIR test) and a comprehensive neuropsychological test battery. Participants also complete questionnaires concerning subjective cognitive complaints, quality of life and general acceptance of virtual reality technology. Functional capacity is assessed using a clinician-rated interview and a performance-based assessment. For participants with mood disorders, mood symptoms are rated with the Hamilton Depression Rating Scale (HDRS-17) and Young Mania Rating Scale (YMRS). For participants with psychosis spectrum disorders, positive and negative symptoms are rated with the Scale for the Assessement of Positive symptoms (SAPS) and Brief Negative Symptom Scale (BNSS), respectively. Finally, sleep quantity and quality in the past 3 days is recorded. Later the same day an fMRI scan is carried out encompassing a spatial working memory N-back task, a word encoding paradigm in which participants must encode and subsequently recognize words of typical household items, a resting state, and a structural scan. On day 2, participants' daily life functional capacity is assessed with The Assessement of Motor and Process Skills (AMPS) by an AMPS-certified occupational therapist in a standardized test kitchen.

The virtual reality cognition test, neuropsychological assessments, questionnaires, clinical symptom ratings, assessements of functional capacity (including AMPS) and fMRI scan are repeated within 2 weeks of treatment completion (primary outcome assessement time). All assessments except for the fMRI scan are repeated again 3 months after treatment completion to assess durability.

Participants are randomized upon full completion of the baseline assessement with allocation being carried out using the automated randomization module in the online Research Electronic Data Capture (REDcap) system based on an uploaded blocked randomization list stratified by age (< or ≥ 35 years) and diagnosis (mood disorders v. psychosis spectrum disorder)

ELIGIBILITY:
Inclusion Criteria:

* Fluent Danish skills
* Meet the International Classification of Diseases 10th edition (ICD-10) diagnosis of unipolar disorder, bipolar disorder (types I and II) or a psychosis spectrum disorder (i.e. F20-F29) confirmed using the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview
* Patients must have objective and subjective cognitive impairment at the time of inclusion. Objective cognitive impairment is defined a total score on the Screen for Cognitive Impairment in Psychiatry - Danish version (SCIP-D) ≥ 0.5 standard deviations (SD) below the expected total score based on age, education, and gender or as a score ≥ 0.5 SD below the expected score on a minimum of two out of the five subtests (verbal learning test - immediate, working memory test, verbal fluency test, verbal learning, test - delayed, and processing speed test). Subjective cognitive impairment is defined as a score ≥ 14 on the Cognitive Complaints in Bipolar Disorder Rating Scale (COBRA).

Exclusion Criteria:

* Current drug or substance abuse
* A daily use of benzodiazepines >22.5 mg oxazepam or >7.5 mg diazepam (cutoffs for doses with limited cognitive side effects)
* Comorbid neurological disorder
* Previous serious head trauma
* Dyslexia
* Pregnancy
* Claustrophobia (fMRI scan)
* Having a pacemaker or other metal implants inside the body (fMRI scan)
* Having had electroconvulsive therapy in the 3 months prior to inclusion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Cognition Assessement in Virtual Reality (CAVIR) test: cognitive composite score | Baseline, treatment completion (primary outcome assessement time point) and 3-months follow-up
  The primary outcome measure is a broad cognitive composite score spanning all five subtasks on a novel virtual reality test of daily-life cognitive functions, the Cognition Assessement in Virtual Reality (CAVIR) test. The CAVIR test is a self-administered 360º immersive VR test in a kitchen, where the participant's abilities to plan and prepare a meal are assessed. The test has a duration of 15 minutes and involves five subtasks probing verbal memory, executive functions, processing speed, working memory and sustained attention, respectively. The cognitive composite score is calculated by averaging the z-transformed scores on the five CAVIR subtasks. No score range. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Rey Auditory Verbal Learning Test (RAVLT): verbal learning and memory domain composite score | Baseline, treatment completion and 3-months follow-up
  A domain composite of 'verbal learning and memory' comprising the following subtests on the Rays Verbal Learning (RAVLT) Test: RAVLT total recall lists I-V, RAVLT immediate recall, RAVLT delayed recall. Score range 0-120. Higher scores mean a better outcome
Assessement of Motor and Process skills (AMPS) | Baseline, treatment completion and 3-months follow-up
  A recommended measure of functioning (i.e. Activity of Daily Living) in individuals with psychiatric illness and cognitive impairment conducted by an AMPS-certificated occupational therapist a standardized test apartment. During an AMPS-evaluation, two domains of performance are evaluated: ADL motor skills (16 items) and ADL process skills (20 items). Scoring of the AMPS assessment is conducted using t available software Occupational Therapy Assessment Package (OTAP) reporting software. OTAP is based on a many-faceted Rasch measurement model making it possible to convert ordinal raw scores into overall linear ADL motor and process ability measures adjusted for severity of the task, skill item difficulty, and rater severity (determined based on rater calibration). A clinically relevant difference has been determined as ≥0.3 logit on the ADL motor or process ability scales. Higher scores mean a better outcome.

OTHER OUTCOMES:
One Touch Stocking of Cambridge | Baseline, treatment completion and 3-months follow-up
  A computerised neuropsychological test assessing executive function. Score range 0-15. Higher scores mean a better outcome
Spatial Working Memory test | Baseline, treatment completion and 3-months follow-up
  A computerised neuropsychological test assessing spatial working memory. Score range 2-14. Higher scores mean a better outcome.
Rapid Visual Information Processing | Baseline, treatment completion and 3-months follow-up
  A computerised neuropsychological test assessing sustained attention. Score range 0-1. Higher scores mean a better outcome.
Wechsler Adult Intelligence Scale Third edition (WAIS-III) letter-number sequencing | Baseline, treatment completion and 3-months follow-up
  Neuropsychological test assessing executive function. Score range 0-21. Higher scores mean a better outcome.
Repeatable Battery of the Assessment of Neuropsychological Status (RBANS) Digit Span | Baseline, treatment completion and 3-months follow-up
  Neuropsychological test assessing attention. Score range 0-16. Higher scores mean a better outcome.
Repeatable Battery of the Assessment of Neuropsychological Status (RBANS) Coding | Baseline, treatment completion and 3-months follow-up
  Neuropsychological test assessing processing speed. Score range 0-89. Higher scores mean a better outcome.
Verbal Fluency with the letter "D" and "S" | Baseline, treatment completion and 3-months follow-up
  Neuropsychological test assessing executive function. No score range. Higher scores mean a better outcome.
Trail Making Test A | Baseline, treatment completion and 3-months follow-up
  Neuropsychological test assessing attention. Scored as time to complete. A higher time means a worse outcome.
Trail Making Test B | Baseline, treatment completion and 3-months follow-up
  Neuropsychological test assessing executive function. Scored as time to complete. A higher time means a worse outcome.
Brief University of California, San Diego Performance-Based Skills Assessment-B (UPSA-B) | Baseline, treatment completion and 3-months follow-up
  Objective assessment of level of functioning. Score range 0-100. Higher scores mean a better outcome.
Wisconsin Card Sorting Task | Baseline, treatment completion and 3-months follow-up
  Computerized neuropsychological test assessing executive function. No score range. Higher scores mean a worse outcome.
Functional Assessment Short Test | Baseline, treatment completion and 3-months follow-up
  Observer-based rating of level of functioning. Score range 0-72. Higher scores mean a worse outcome.
Cognitive Complaints in Bipolar Disorder Rating Assessement (COBRA) | Baseline, treatment completion and 3-months follow-up
  Questionnaire on subjective cognitive complaints. Score range 0-48. Higher scores mean a worse outcome.
World Health Organization Quality of Life (WHOQOL-BREF) | Baseline, treatment completion and 3-months follow-up
  Questionnaire on quality of life. Score range 26-130. Higher scores mean a better outcome.
Cognitive Difficulties in Everyday Life (CODEL) | Baseline, treatment completion and 3-months follow-up
  Questionnaire on subjective cognitive complaints. Score range 0-48. Higher scores mean a worse outcome
Perceived Competence Scale (PCS) | Baseline, treatment completion and 3-months follow-up
  Questionnaire on self-efficacy. Score range 0-49. Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kamilla Woznica Miskowiak, DMSc, DPhil, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Neurocognition and Emotion in Affective Disorders (NEAD) Centre, Copenhagen Affective Disorder Research Centre (CADIC), Psychiatric Centre Copenhagen, Frederiksberg hospital, Frederiksberg, Capital Region of Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miskowiak KW, Jespersen AE, Kessing LV, Aggestrup AS, Glenthoj LB, Nordentoft M, Ott CV, Lumbye A. Cognition Assessment in Virtual Reality: Validity and feasibility of a novel virtual reality test for real-life cognitive functions in mood disorders and psychosis spectrum disorders. J Psychiatr Res. 2022 Jan;145:182-189. doi: 10.1016/j.jpsychires.2021.12.002. Epub 2021 Dec 12. PMID 34923359
- [Derived] Jespersen AE, Lumbye A, Vinberg M, Glenthoj L, Nordentoft M, Waehrens EE, Knudsen GM, Makransky G, Miskowiak KW. Effect of immersive virtual reality-based cognitive remediation in patients with mood or psychosis spectrum disorders: study protocol for a randomized, controlled, double-blinded trial. Trials. 2024 Jan 24;25(1):82. doi: 10.1186/s13063-024-07910-7. PMID 38268043